CLINICAL TRIAL: NCT01153945
Title: Association Between Cancer Cells and Normal Vs. Low Levels of Thyroid Hormones in the Serum
Brief Title: Association Between Cancer Cells and Normal Versus (Vs.) Low Levels of Thyroid Hormones in the Serum
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor stopped the study.
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 097-2010
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2011-08

CONDITIONS: Thyroid Cancer
Keywords: Hypothyroid and non hypothyroid
MeSH Terms: conditions — Thyroid Neoplasms; Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hypothyroid
- Non hypothyroid
- Healthy subjects

SUMMARY:
Much experimental data has suggested that thyroid hormones (T3 and T4) may modulate neoplastic cells and that T3/T4 deprivation may remove this stimulus. It is now well established that T3/T4 affects cell division/angiogenesis through binding to integrin avb3, commonly over-expressed on many cancer cells. In the experimental settings, mimicking hypothyroidism in the cells is a difficult task. Currently, the use of charcoal stripped serum is used. Using this method, the serum is stripped not only from T3 and T4, as intended, but also from central and important cytokines and growth factor. This leads to a reduced rate of cancer cell proliferation and thus, does not reflect the natural environment in which cancer cells residue under hypothyroid conditions.

The investigators aim to characterize and establish the effects of serum from hypothyroid patients on the proliferation/viability of a variety of cancer cell models.

ELIGIBILITY:
Inclusion Criteria:

* Hypothyroid state

Exclusion Criteria:

* Non hypothyroid state

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid cancer patients before/after radioactive iodine total body scan or treatment admitted to the Endocrinology Institute, Meir Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nabriski, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel